CLINICAL TRIAL: NCT06149286
Title: A Phase 3, Open Label, Randomized Study to Compare the Efficacy and Safety of Odronextamab (REGN1979), an Anti-CD20 x Anti-CD3 Bispecific Antibody, in Combination With Lenalidomide Versus Rituximab in Combination With Lenalidomide in Relapsed/Refractory Participants With Follicular Lymphoma and Marginal Zone Lymphoma (OLYMPIA-5)
Brief Title: A Trial to Find Out if Odronextamab Combined With Lenalidomide is Safe and Works Better Than Rituximab Combined With Lenalidomide in Adult Participants With Follicular Lymphoma and Marginal Zone Lymphoma
Acronym: OLYMPIA-5
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1979-ONC-22102; 2022-503092-28-00 (EU CTIS Number)
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Follicular Lymphoma; Relapsed/Refractory Marginal Zone Lymphoma (R/R MZL)
Keywords: Relapsed/Refractory Follicular Lymphoma; Relapsed/Refractory Marginal Zone Lymphoma; Non-Hodgkin lymphomas; Indolent lymphomas; Odronextamab
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence; Lymphoma, B-Cell, Marginal Zone | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Odronextamab+Lenalidomide (Experimental): In part 1 (safety run-in), participants with R/R indolent lymphoma (FL and MZL), will receive odronextamab in combination with lenalidomide.
  In part 2, 1:1 randomized participants with R/R indolent lymphoma (FL/MZL), will receive odronextamab in combination with lenalidomide.
  Interventions: Drug: Odronextamab; Drug: Lenalidomide
- Rituximab+Lenalidomide (Experimental): In part 2 only, 1:1 randomized participants with R/R lymphoma (FL and ML), will receive rituximab in combination with lenalidomide (R2) followed by lenalidomide monotherapy.
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Odronextamab — Administered per the protocol
  Other Names: REGN1979; Ordspono
  Arms: Odronextamab+Lenalidomide
Drug: Lenalidomide — Administered per the protocol
  Other Names: REVLIMID
Drug: Rituximab — Administered per the protocol
  Other Names: Rituxan
  Arms: Rituximab+Lenalidomide

SUMMARY:
This study is researching an experimental drug called odronextamab (referred to as study drug), in combination with lenalidomide. The study is focused on participants who have one of two types of cancer: follicular lymphoma (FL) or marginal zone lymphoma (MZL) that has come back after treatment (called "relapsed"), or did not respond to treatment (called "refractory"). FL and MZL are subtypes of Non-Hodgkin 's lymphoma (NHL).

This study will be made up of two parts (Part 1 not randomized, Part 2 randomized - controlled).

The aim of Part 1 of the study is to see how safe and tolerable the study drug is when used in combination with lenalidomide, in participants with FL or MZL, and to determine the dose of the study drug to be used in Part 2 of this study. This combination is considered "first-in-human" as it has not been tested as a combination treatment in humans before.

The aim of Part 2, of the study is to assess how well the combination of the study drug and lenalidomide works compared to the combination of rituximab (called "the comparator drug") and lenalidomide. The combination of comparator drug and lenalidomide is the current standard-of-care treatment for relapsed/refractory FL and/or MZL. Standard-of-care means the usual medication expected and used when receiving treatment for a condition.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug in combination with lenalidomide
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)
* The impact from the study drug on quality-of-life and ability to complete routine daily activities

ELIGIBILITY:
Key Inclusion Criteria:

1. Local histologic confirmation of FL grade 1-3a or MZL (nodal, splenic, or extra nodal MZL) as assessed by the investigator, as described in the protocol.
2. Must have refractory disease or relapsed after at least 1 prior line (with a duration of at least 2 cycles) of systemic chemo-immunotherapy or immunotherapy. Prior systemic therapy should have included at least one anti-Cluster of Differentiation 20 (CD20) monoclonal antibody and participant should meet indication for treatment, as described in the protocol.
3. Have measurable disease on cross sectional imaging documented by diagnostic Computed Tomography [CT], or Magnetic Resonance Imaging [MRI] imaging, as described in the protocol.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Adequate hematologic and organ function, as described in the protocol.
6. All study participants must:

   1. Have an understanding that lenalidomide could have a potential teratogenic risk.
   2. Agree to abstain from donating blood while taking study drug therapy and for 28 days after discontinuation of lenalidomide.
   3. Agree not to share study medication with another person.
   4. Agree to be counseled about pregnancy precautions and risk of fetal exposure associated with lenalidomide.

Key Exclusion Criteria:

1. Primary Central Nervous System (CNS) lymphoma or known involvement (either current or prior history of CNS involvement) by non-primary CNS NHL, as described in the protocol.
2. Participants with current or past histological evidence of high-grade or diffuse large B-cell lymphoma, or any histology other than FL grade 1-3a or MZL.
3. History of or current relevant CNS pathology, as described in the protocol.
4. A malignancy other than NHL (inclusion diagnosis) unless the participant is adequately and definitively treated and is cancer free for at least 3 years, with the exception of localized prostate cancer treated with hormone therapy or local radiotherapy (ie, pellets), cervical carcinoma in situ, breast cancer in situ, or nonmelanoma skin cancer that was definitively treated.
5. Any other significant active disease or medical condition that could interfere with the conduct of the study or put the participant at significant risk, as described in the protocol.
6. Allergy/hypersensitivity to study drugs or excipients. as described in the protocol.
7. Active infection as defined in the protocol.

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2029-01-23 (Estimated); Study Completion 2029-01-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) for odronextamab in combination with lenalidomide | Up to 35 days
  Part 1
Incidence of Treatment Emergent Adverse Events (TEAEs) for odronextamab in combination with lenalidomide | Up to 2 years
  Part 1
Severity of TEAEs for odronextamab in combination with lenalidomide | Up to 2 years
  Part 1
Progression-Free Survival (PFS) as assessed by Independent Central Review (ICR) in participants with R/R FL and participants with indolent lymphoma | Up to 5 years
  Part 2

SECONDARY OUTCOMES:
Odronextamab concentrations in serum | Up to 30 months
  Part 1 and Part 2
Incidence of Anti-drug Antibodies (ADA) to odronextamab | Up to 30 months
  Part 1 and Part 2
Magnitude of ADAs to odronextamab | Up to 30 months
  Part 1 and Part 2
Best Overall Response (BOR) as assessed by investigator review | Up to 30 months
  Part 1 and Part 2
Duration of Response (DOR) as assessed by investigator review | Up to 5 years
  Part 1 and Part 2
PFS as assessed by investigator review | Up to 5 years
  Part 1 and Part 2
Complete Response (CR) as assessed by ICR | Up to 30 months
  Part 2
BOR as assessed by ICR | Up to 30 months
  Part 2
Overall Survival (OS) | Up to 5 years
  Part 2
Event Free Survival (EFS) as assessed by ICR | Up to 5 years
  Part 2
EFS as assessed by local investigator review | Up to 5 years
  Part 2
DOR as assessed by ICR | Up to 5 years
  Part 2
Time To Next anti-lymphoma Treatment (TTNT) | Up to 5 years
  Part 2
Incidence of TEAEs for odronextamab in combination with lenalidomide versus R2 | Up to 2 years
  Part 2
Severity of TEAEs for odronextamab in combination with lenalidomide versus R2 | Up to 2 years
  Part 2
Overall change in patient reported outcomes (PROs) as measured by scores of European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire (EORTC QLQC30) | Up to 5 years
  Part 2 The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a global health status (GHS)/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status/QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
Overall change in PROs as measured by scores of Functional Assessment of Cancer Therapy-Lymphoma Subscale (FACT-LymS) | Up to 5 years
  Part 2 The FACT-Lym lymphoma subscale (LymS) includes 15 items to assess NHL-related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). Higher scores are associated with a worse quality of life.
Overall change in PROs as measured by scores of EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L) | Up to 5 years
  Part 2 The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: "no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems". The EQ VAS records the participant's self-rated health on a vertical visual analogue scale where the endpoints are labeled "Best imaginable health state" and "Worst imaginable health state".
Change from first assessment in Patient Global Impression on Severity (PGIS) | Up to 5 years
  Part 2 The PGIS includes a single-item to assess how a patient perceives the overall severity of cancer symptoms over the past 7 days. Patients will choose the response that best describes the severity of their overall cancer symptoms with options on a 5-point scale ranging from 1 (No symptoms) to 4 (Very Severe).
Change from first assessment in Patient Global Impression on Change (PGIC) | Up to 5 years
  Part 2 The PGIC item includes a single-item to assess how a patient perceives their overall change in health status since the start of study treatment. Patients will choose from response options on a 7-point scale ranging from 1 (Much Better) to 7 (Much worse); 1- Much Better, 2-Moderately Better, 3-A Little Better, 4-About the Same, 5-A Little Worse, 6-Moderately Worse, 7-Much Worse.
Change from first assessment in the Global Population item 5 (GP5) items of the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire | Up to 5 years
  Part 2 A single item (GP5) of the validated FACT-G questionnaire will be used to assess from the participant perspective the overall impact of treatment side-effect. The question item is on a 5-point scale ranging from "not at all" (0) to "very much" (4).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (167):
- United States (8):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Boca Raton Clinical Research (BRCR) Global, Plantation, Florida
  - Indiana University and Comprehensive Cancer Center, Indianapolis, Indiana
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Dartmouth Cancer Center, Lebanon, New Hampshire
  - Stony Brook University Hospital, Stony Brook, New York
  - Clinical Research Alliance Inc, Westbury, New York
  - Prohealth Care Inc, Waukesha, Wisconsin
- Australia (5):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Epworth Freemasons, East Melbourne, Victoria
- Austria (4):
  - Ordensklinikum Linz, Linz, Osterreich
  - Kepler University Hospital, Linz, Upper Austria
  - Medical University Vienna, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (5):
  - Centre Hospitalier Universitaire at Universite Catholique de Louvain Namur, Yvoir, Namur
  - Universitair Ziekenhuis (UZ) Gent/ Ghent University Hospital, Ghent, Oost-Vlaanderen
  - Algemeen Ziekenhuis AZ Delta, Roeselare, West-Vlaanderen
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Institut Jules Bordet, Brussels
- Brazil (10):
  - Hospital Sao Rafael, Salvador, Estado de Bahia
  - Hospital Sirio Libanes Brasilia, Brasília, Federal District
  - Uopeccan Hospital do Cancer de Cascavel, Cascavel, Paraná
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado, Porto Alegre, Rio Grande do Sul
  - Amaral Carvalho Hospital, Jaú, São Paulo
  - Instituto Nacional de Cancer Jose Alencar Gomes da Silva, Rio de Janeiro
  - Hospital Sirio Libanes, São Paulo
  - A Beneficencia Portuguesa de Sao Paulo, Oncology House, São Paulo
- Czechia (4):
  - University Hospital Hradec Kralove, Hradec Králové, East Bohemia
  - Fakultni Nemocnice Brno, Brno
  - University Hospital Kralovske Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- France (17):
  - Institut Paoli-Calmettes, Marseille, Bouches Du Rhone
  - CHU de Rennes, Rennes, Brittany Region
  - Centre Hospitalier Regional Universitaire de Tours, Tours, Centre-Val de Loire
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux, Gironde
  - Centre Francois Magendie, Pessac, Gironde
  - Hopital Saint Vincent-de-Paul, Lille, Nord
  - Centre Henri Becquerel, Rouen, Normandy
  - Nantes University Hospital, Nantes, Pays de la Loire Region
  - Centre Hospitalier Metropole Savoie, Chambéry, Savoie
  - Centre Hospitalier d'Avignon, Avignon
  - Centre Hospitalier Universitaire (CHU) Montpellier, Montpellier
  - Hopital Saint Louis, Paris
  - Assistance Publique-Hopitaux de Paris (AP-HP), Paris
  - Institut Curie, Saint-Cloud
  - Hopital Victor Dupouy Argenteuil, Argenteuil, Île-de-France Region
  - Avicenne Hospital, Bobigny, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region
- Germany (7):
  - Stauferklinikum, Mutlangen, Baden-Wurttemberg
  - Robert-Bosch-Krankenhaus, Stuttgart, Baden-Wurttemberg
  - LMU Klinikum, Munich, Bavaria
  - Clinic Frankfurt (Oder), Frankfurt am Main, Hesse
  - Universitatsmedizin der Johannes-Gutenberg Universitat Mainz, Mainz, Rhineland-Palatinate
  - Stadtisches Krankenhaus Kiel, Kiel
  - MVZ fuer Haematologie und Onkologie Rhein-Kreis GmbH, Neuss
- Israel (7):
  - Assuta Ashdod Medical Center, Ashdod
  - Hadassah Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Medical Centers, Tel Aviv
- Italy (18):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli-Cesena
  - Ospedale Policlinico San Martino IRCCS, Genoa, Genova
  - S Gerardo Hospital, Monza, Monza E Brianza
  - A.O.U. Citta della Salute e della Scienza di Torino, Turin, Piedmont
  - Centro Di Riferimento Oncologico (CRO), Aviano, National Cancer Institute, Aviano, Pordenone
  - Candiolo Cancer Institute, FPO, IRCCS, Candiolo, Torino
  - University of Bologna Dipartimento di Medicina Specialistica Diagnostica e Sperimentale, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - ASST Grande Ospedale Metropolitano Niguarda - Main Address, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Istituto Europeo di Oncologia, Milan
  - A.O.U. di Modena, Modena
  - Federico II University, Napoli
  - AOU Maggiore della Carita, Novara
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera di Perugia, Perugia
  - Ospedale Santa Maria delle Croci, Ravenna
  - Santa Maria della Misericordia, Udine
- Malaysia (5):
  - Hospital Sultanah Aminah Jhor Bahru, Johor Bahru, Johor
  - University of Malaya Medical Centre, Kuala Lumpur, Negeri / Wilayah Persekutuan
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Hospital Ampang, Ampang, Selangor
  - Subang Jaya Medical Center, Subang Jaya, Selangor
- Poland (11):
  - Specjalistyczny Szpital im A. Sokolowskiego w Walbrzychu, Wałbrzych, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny, Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny Nr 4 w Lublinie, Centrum Innowacyjnych Terapii, Lublin, Lublin Voivodeship
  - Pratia MCM Krakow, Krakow, Malopolska
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Pratia Poznan Medical Center, Poznan, Wielkopolska
  - Aidport, Skorzewo, Wielkopolska
  - Szpital Uniwersytecki Nr2 Bydgoszcz, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. Mikolaja Kopernika w Lodzi (Copernicus Memorial Hospital), Lodz
  - Narodowy Instytut Onkologii, Warsaw
- South Korea (13):
  - St. Vincents Hospital - The Catholic University of Korea, Suwon, Gyeonggi-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk
  - Gachon University Gil Medical Center, Incheon, Namdong-Gu
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Yeyungnam University Medical Center, Daegu
  - Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Yeouido St. Marys Hospital, Seoul
  - Seoul St Marys Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (18):
  - University Hospital of Santiago de Compostela, Santiago de Compostela, A Coruna
  - Son Espases University Hospital, Palma, Balearic Islands
  - Institut Catala d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - University Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Virgen De Las Nieves De Granada, Granada
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital Universitario12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - University Hospital Virgen del Rocio, Seville
  - Instituto Valenciano de Oncologia, Valencia
  - University Hospital Doctor Peset, Valencia
- Taiwan (12):
  - Chang Gung Medical Foundation Chia Yi Branch, Buzi, Chiayi County
  - Changhua Christian Hospital, Changhua
  - Show Chwan Memorial Hospital, Changhua
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan
- Thailand (3):
  - Chulalongkorn University, Bangkok, Krung Thep Maha Nakhon [Bangko]
  - Sriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
- Turkey (Türkiye) (11):
  - Ankara University Faculty of Medicine, Mamak, Ankara
  - Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Yenimahalle, Ankara
  - Gazi University, Ankara, Central Anatolia
  - VM Medical Park Mersin Hospital, Mezitli, Mersin
  - Tekirdag Namik Kemal University Hospital, Tekirdağ, Suleymanpasa
  - Istanbul University, Istanbul Medical Faculty, Istanbul
  - Ege University, Izmir
  - Dokuz Eylul University, Izmir
  - Sakarya University Medical Faculty, Sakarya
  - Ondokuz Mayıs University, Samsun
  - Zonguldak Bulent Ecevit University, Zonguldak
- United Kingdom (9):
  - Royal Cornwall Hospital NHS Trust, Truro, Cornwall
  - Derriford Hospital and the Royal Eye Infirmary, Plymouth, Devon
  - University Hospitals Dorset, Bournemouth, Dorset
  - Salisbury Foundation Trust, Salisbury, Hampshire
  - The Hillingdon Hospital, Uxbridge, Middlesex
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth
  - Barking, Havering and Redbridge University Hospitals NHS Trust, Romford
  - South Warwickshire NHS Foundation Trust, Warwick

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: OLYMPIA — https://olympiastudies.com/en-us